CLINICAL TRIAL: NCT05226091
Title: TRial to Assess Implementation of New Research in a Primary Care Setting (TRAINS): a Pragmatic Cluster Randomised Controlled Trial of an Educational Intervention to Promote Asthma Prescription Uptake in General Practitioner Practices
Brief Title: Trial to Assess Implementation of New Research in a Primary Care Setting (TRAINS)
Acronym: (TRAINS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 174770
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2021-12

CONDITIONS: General Practice (GP), Primary Care Settings
MeSH Terms: interventions — College Fraternities and Sororities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): GP practices randomised to the intervention will receive a mail and email about the result of the PLEASANT study and advising them to implement the study findings.
  Interventions: Behavioral: Letter
- Usual care arm (No Intervention): GP practices randomised to control will not receive either mail or email and they will continue with usual care.

INTERVENTIONS:
Behavioral: Letter — Selected GP practices currently registered with CPRD will receive correspondence by both email and mail informing them about the result of the PLEASANT study and advising them how to implement what has been learnt. Included in the mailing would be a suggested letter and SMS text.
  Arms: Intervention arm

SUMMARY:
In England and Wales, unscheduled care for school-aged children with asthma significantly increases after their return to school in September, a trend linked with decreased asthma preventer prescriptions during the summer holidays. The PLEASANT study found that a reminder letter from GPs to parents of children with asthma led to a 30% increase in prescription uptake during August and reduced unscheduled medical visits from September to December.

The TRAINS trial will now assess if informing GPs of PLEASANT findings would lead to its implementation. This pragmatic cluster randomised implementation trial will use routine data from Clinical Practice Research Datalink (CPRD).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of practices Practices inclusion criteria

  1- General practices who are currently contributing part of the CPRD in England.
* Inclusion criteria of children with asthma

Inclusion criteria for the data extraction from CPRD:

1- School-aged children with asthma aged between 4 to 16 years old as of 1st September 2021 with a coded diagnosis of asthma who have been prescribed asthma medication in the last 12 months.

Exclusion Criteria:

* Practice exclusion criteria:

  1. General practices that are not in England.
  2. General practices that are not included in the CPRD.
  3. Practices that cease to be part of the CPRD during the intervention time without contributing to the primary outcome.
  4. Practices that merge during the intervention (where the merging practices were in different study arms).
* Exclusion criteria of children with asthma:

  1. School-aged children with asthma under 4 and over 16 years old as of 1st September 2021.
  2. Children with no asthma diagnosis
  3. Children with asthma who have not received a prescription for asthma medication. in the last 12 months

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1389 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion of children with asthma who have a prescription for an asthma preventer medication from 1st August 2021 to 30th September 2021. | 8 weeks
  prescription uptake of asthma preventer medication for children with asthma.

SECONDARY OUTCOMES:
The number of asthma preventer medication prescriptions per School-aged child with asthma patient from 1st August 2021 to 30th September 2021. | 8 weeks
  preventer medication prescriptions per School-aged child with asthma patient.
The number of prescription uptake of asthma preventer medication per patient in the month of August 2021. | 4 weeks
  prescription uptake of asthma preventer medication per patient.
The number of prescription uptake of asthma preventer medication per patient in the month of September 2021 | 4 weeks
  prescription uptake of asthma preventer medication per patient.
The proportion of children who have a prescription for asthma preventer medication per patient in the month of August 2021. | 4 weeks
  The proportion of children who have a prescription for asthma preventer medication per patient
The proportion of children who have a prescription for asthma preventer medication per patient in the month of September 2021. | 4 weeks
  children who have a prescription for asthma preventer medication per patient
The number of prescription uptake of asthma preventer medication in the 6 months following the intervention 1st July 2021. | 6 months
  The number of prescription uptake of asthma preventer medication
The proportion of patients with unscheduled medical contact from 1st September 2021 to 30th December 2021 and the individual months of 1st September 2021 to 31st December 2021. | 4 months
  The proportion of patients with unscheduled medical contact
The number of unscheduled medical contact per patient from 1st September 2021 to 31th December 2021 and the individual months from 1st September 2021 to 31st December 2021. | 4 months and each one of them
  The number of unscheduled medical contact per patient
The proportion of patients who have a medical contact (either unscheduled and scheduled) from 1st September 2021 to 30th December 2021 and the individual months from 1st September 2021 to 31st December 2021. | 4 months and each one of them
  The proportion of patients who have a medical contact (either unscheduled and scheduled)
The total number of medical contact (either unscheduled and scheduled) per patient in the period 1st September 2021 to 30th December 2021 and the individual months of 1st September 2021 to 31st December 2021. | 4 months and each one of them
  The total number of medical contact (either unscheduled and scheduled) per patient
The proportion of patients who have an unscheduled medical contact in the period 1st September 2021 to 30th December 2021 and the individual months of 1st September 2021 to 30th December 2021 associated with a respiratory diagnosis. | 4 months and each one of them
  The proportion of patients who have an unscheduled medical contact associated with a respiratory diagnosis.
The number of unscheduled medical contacts per patient and from 1st September 2021 to 30th December 2021 and the individual months of 1st September 2021 to 31st December 2021associated with a respiratory diagnosis. | 4 months and each one of them
  The number of unscheduled medical contacts per patient associated with a respiratory diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Julious, PhD, Study Director — University of Sheffield
Locations (1):
- The University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alyami RA, Simpson R, Oliver P, Campbell R, Julious SA. A letter intervention to GPs practices to promoting prescription uptake in school-age children with asthma during summer holidays (TRAINS study): a pragmatic cluster randomised controlled trial. NPJ Prim Care Respir Med. 2026 Feb 10;36(1):12. doi: 10.1038/s41533-025-00475-1. PMID 41667505
- [Derived] Alyami RA, Simpson R, Oliver P, Julious SA. Evaluation of the impact of letters to GP practices to promote asthma prescription uptake in school-age children during summer (TRAINS study): a pragmatic cluster-randomised controlled trial. Lancet. 2023 Nov;402 Suppl 1:S22. doi: 10.1016/S0140-6736(23)02089-5. PMID 37997062
- [Derived] Alyami RA, Simpson R, Oliver P, Julious SA. TRial to Assess Implementation of New research in a primary care Setting (TRAINS): study protocol for a pragmatic cluster randomised controlled trial of an educational intervention to promote asthma prescription uptake in general practitioner practices. Trials. 2022 Nov 17;23(1):947. doi: 10.1186/s13063-022-06864-y. PMID 36397087
- See also: PLEASANR Trial — http://www.sheffield.ac.uk/scharr/research/centres/ctru/pleasant
- See also: Rami's Page — http://www.sheffield.ac.uk/scharr/people/pgr-students/rami-ali-h-alyami